CLINICAL TRIAL: NCT03459911
Title: A Randomized, Open-label, Single-dose, Two-treatment, Two-sequence, Two-period, Crossover Bioequivalence Study of Test Losartan Potassium Tablets (Containing Losartan Potassium 100 mg) of Pharmtechnology LLC, Republic of Belarus With Reference Cozaar® (Containing Losartan Potassium 100 mg) of "Merck Sharpe & Dohme B.V.", Haarlem, the Netherlands in Normal, Healthy, Adult, Human Subjects Under Fasting Conditions
Brief Title: A Bioequivalence Study of Losartan Potassium Tablets (Containing Losartan Potassium 100 mg) in Normal, Healthy, Adults Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pharmtechnology LLC (Industry)
Collaborators: Reliance Life Sciences Private Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: RLS/1117/046
Record Dates: First submitted 2018-02-27; First posted 2018-03-09 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-06

CONDITIONS: Healthy
Keywords: Bioequivalence
MeSH Terms: interventions — Losartan; Tablets

STUDY DESIGN:
Masking Description: This study is an open label study; the subjects and the investigator will not be blinded towards the identity of the investigational products. However, analysts will be blinded towards identity of investigational product administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Losartan potassium 100 mg Tablets (Experimental): Losartan potassium is the test product. In period 1 and period 2, 33 of 66 subjects will be given single oral dose (1 x 100 mg) of Losartan potassium.
  Interventions: Drug: Losartan potassium 100mg
- Cozaar® (Losartan potassium)100 mg Tablets (Active Comparator): Cozaar® (Losartan potassium) is the reference product. In period 1 and period 2, 33 of 66 subjects will be given single oral dose (1 x 100 mg) of Cozaar®.
  Interventions: Drug: Cozaar 100mg Tablet

INTERVENTIONS:
Drug: Cozaar 100mg Tablet — Cozaar® ( Losartan potassium) 100 mg Tablets(Merck Sharpe & Dohme B.V. , Haarlem, the Netherlands)
  Arms: Cozaar® (Losartan potassium)100 mg Tablets
Drug: Losartan potassium 100mg — Losartan potassium 100 mg Tablets ( Pharmtechnology LLC, Republic of Belarus)
  Arms: Losartan potassium 100 mg Tablets

SUMMARY:
To demonstrate bioequivalence of single dose test formulation of Losartan potassium tablets (containing Losartan potassium 100 mg) of Pharmtechnology LLC, Republic of Belarus with reference Cozaar® (containing Losartan potassium 100 mg) of "Merck Sharpe & Dohme B.V.", Haarlem, the Netherlands in normal, healthy, adult, human subjects under fasting conditions.To monitor adverse events and ensure the safety

DETAILED DESCRIPTION:
Total 66 normal healthy adult subjects will be enrolled in the study. Subjects will be administered either the Test or the Reference Product with 200 mL of water in each period as per the randomization schedule. Subjects will fast for at least 10 hours prior to administration of the study drugs and for four (4) hours after administration of the study drugs during each study period. Standardized meals will be provided in each study period. Water will not be accessible to the subjects 1 hour to administration of the study drugs and 1 hour after administration of the study drugs in each period. A total of 29 blood samples will be withdrawn for pharmacokinetic profiling during each study period. The plasma concentrations of losartan and its carboxylic acid metabolite will be measured by a validated LC-MS/MS analytical method. ANOVA will be performed on log transformed pharmacokinetic parameters Cmax, AUC0-t, AUC0-∞, and 90% confidence interval will be constructed for the ratio of geometric least square mean of the Test and Reference products, obtained from the log-transformed data. Bioequivalence will be concluded if the ratio estimate as well as its 90% confidence interval, both falls within the acceptable range of 80.00% to 125.00% for Cmax, AUC0-t.

ELIGIBILITY:
Inclusion Criteria:

The following criteria should be checked at the time of study entry. If any does not apply at the time of study entry, the subject must not be included in the study:

1. Healthy adult human subjects, aged between 18 to 45 years (both inclusive).
2. Subjects with Body Mass Index (BMI) 18.5 to 24.9 kg/m2
3. Subjects able and willing to comply with the protocol requirements.
4. Subjects should not have any medical history of significant diseases.
5. If subject is a female and is

   * of child bearing potential, she should be practicing an acceptable method of birth control for the duration of the study as suggested by the investigator, such as a combination of male condom with either cap, diaphragm or sponge with spermicide (double barrier method), intrauterine device (IUD), or abstinence.

   OR
   * surgically sterile, bilateral tubal ligation done at least 6 months before the study should be documented.
6. Subjects willing to voluntarily provide written informed consent.
7. Subjects willing to undergo pre- and post-study physical examinations and laboratory investigations.
8. Subjects who are non-smokers based on history.
9. Subjects willing to adhere to the protocol and the following study requirements:

   * Should not consume xanthine containing products, such as coffee, tea, chocolate or soft drinks at least 48 hours prior to dosing (i.e. in-house monitoring and the remaining based on history) until the last sample collection.
   * Should not consume alcohol at least 48 hours prior to dosing (i.e. during in-house monitoring and the remaining based on history) until the last sample collection.
   * Should not consume grapefruit or its products at least 7 days prior to each dosing (i.e. during in-house monitoring and the remaining based on history) and until the last sample collection.
10. Subjects having no clinically significant medical history and no clinically significant abnormalities in general physical examination, laboratory assessments, 12-lead ECG, chest X-Ray or vital signs.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any of these apply at the time of study entry, the subject must not be included in the study:

1. Subjects incapable of understanding the informed consent process.
2. Female subjects with a positive pregnancy test at screening or positive serum β-HCG test (done at check-in of each study periods) or lactating females.
3. Female subjects of childbearing potential who are unwilling or unable to use an appropriate method of contraception as outlined in the inclusion criteria, at least 28 days prior to the first period dosing until the post-study follow-up (i.e. until 7 days from the drug administration in Period II). Use of hormonal contraceptives either oral or implants within 3 months prior to first period dosing will not be acceptable.
4. Subjects with inadequate venous access in their left or right arm to allow the collection of all samples via venous cannula in the study.
5. Subjects with abnormalities in resting heart rate (>100 beats/min or <50 beats/min), blood pressure either hypotensive episode (systolic blood pressure <90 mmHg or diastolic blood pressure <60 mmHg) or hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥90 mmHg), oral temperature (< 95.60F or > 990F) on the screening day.
6. Subjects with history of psychiatric disorders, which are likely to limit the validity of consent to participate in the study, or limit the ability to comply with the protocol requirements.
7. Subjects with any evidence of organ dysfunction or any clinically significant deviation from normal in their physical or clinical evaluation including ECG and X-ray results.
8. Subjects who have taken over the counter or prescribed medications, including any enzyme modifying drugs or any systemic medication within 30 days prior to the start of the clinical period and during the study period.
9. Subjects with a known history of drug hypersensitivity to losartan or any excipients of the formulation.
10. Subjects with a history of alcohol abuse and/or drug abuse or who are found urinary screen test positive for drugs of abuse (Amphetamines, Morphine, Benzodiazepines, Marijuana, Cocaine and Barbiturates) or are found with current alcohol abuse based on alcohol breath test.
11. Subjects diagnosed to be HIV 1 and 2 or Hepatitis B (HBsAg) or Hepatitis C (HCV) virus positive.
12. Subjects with clinically significant abnormal haematological values [haemoglobin (Hb), total white blood cells count (WBC), total red blood cells count (RBC), differential WBC count, platelet count and hematocrit].
13. Subjects with clinically significant abnormal laboratory values for serum creatinine, blood urea nitrogen (BUN), serum aspartate aminotransferase (AST), serum alanine aminotransferase (ALT), serum alkaline phosphatase (ALP), serum bilirubin, serum glucose (fasting), and serum cholesterol.
14. Subjects with clinically significant abnormal urine analysis, defined as the presence of RBC (>5/HPF), pus cells (>5/HPF), epithelial cells (>5/HPF), glucose (positive), ketones (positive), bilirubin (positive) and protein (positive) (unless the clinical investigator considers the deviation to be irrelevant for the purpose of the study).
15. Subjects with a clinically significant past history or current medical condition of:

    1. Pulmonary disorders (COPD and asthma)
    2. Cardiovascular disorders (especially heart blocks, myocardial infarction, congestive heart failure and uncontrolled hypertension)
    3. Neurological disorders (especially epileptic seizures)
    4. GIT disorders (gastrointestinal bleeding, gastric/peptic ulcer)
    5. Renal and/or hepatic disorders
    6. Coagulation disorders
    7. Endocrine disorders (especially diabetes mellitus)
16. Any history of difficulty in donating blood
17. Any clinically significant illness during 3 months before screening.
18. Subjects who participated in any other clinical investigation using experimental drugs or have bled more than 300 mL in the past 3 months

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2018-03-11 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter for losartan | 10 Days
  Peak Plasma Concentration (Cmax)
Pharmacokinetic parameter for losartan | 10 Days
  Area under the plasma concentration versus time curve from time 0 to the last measured concentration (AUC0-t)

SECONDARY OUTCOMES:
Safety and tolerability of investigational products | 17 Days
  Number of adverse events, number of deaths, number of severe adverse events in subjects who have taken at least one dose of investigational products.
Other pharmacokinetic parameters for losartan | 10 Days
  Area under the plasma concentration versus time curve from time 0 to to infinite time(AUC0-∞)
Other pharmacokinetic parameters for losartan | 10 Days
  Time of maximum measured plasma concentration (Tmax)
Other pharmacokinetic parameters for losartan | 10 Days
  Elimination or terminal half-life (T1/2)
Other pharmacokinetic parameters for losartan | 10 Days
  Elimination rate constant (Kel)
Other pharmacokinetic parameters for losartan | 10 Days
  Residual area (AUCresid)

CONTACTS AND LOCATIONS:
Overall Officials: Suresh A Maroli, MD, Principal Investigator — Reliance Life Sciences Pvt. Ltd
Locations (1):
- Clinical Unit, Reliance Life Sciences Pvt. Ltd., Mumbai, Maharashtra, India

IPD SHARING:
Plan to Share IPD: Undecided
The Company may provide the individual participant data after privacy protection on case by case basis.